CLINICAL TRIAL: NCT05068362
Title: Auricular Reconstruction in Microtia by Medpor Implant Following Tissue Expansion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mina Youssef Asham Gendy, Assistant Lecturer of ENT, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AssiutU 5
Record Dates: First submitted 2021-08-23; First posted 2021-10-05 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Microtia
MeSH Terms: conditions — Congenital Microtia

STUDY DESIGN:
Intervention Model Description: Children with microtia
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implant (Other): Use of Medpor implant in auricle reconstruction in microtia
  Interventions: Device: Auricular reconstruction

INTERVENTIONS:
Device: Auricular reconstruction — Medpor implant for treatment of microtia

SUMMARY:
The study involves patients with microtia of certain criteria will undergo tissue expansion by silicone bags in the postauricular region then Medpor implants will be applied undercover of the expanded skin for reconstruction of the auricule instead of the costal cartilage graft

DETAILED DESCRIPTION:
Background :

Autologous multistage rib cartilage technique for auricular reconstruction was firstly introduced by Tanzer in 1959(1) however, such technique had many drawbacks like being a lengthy process consisting of multiple procedures, donor-site morbidity and pain and the possibility of cartilage resorption leading to poor ear projection and loss of auricular definition (2). Tjellström (3) and Korus et al (4) described the osseointegrated implant for auricular reconstruction in traumatic congenital and oncological conditions. It also had disadvantages as the need for long-term commitment of both patient and prosthetic team, high costs of maintenance visits, regular change of the prosthesis every 2 to 5 years and the prosthesis is considered as a foreign body (5). Medpor is a synthetic biocompatible porous polyethylene implant (5) that was used as an alternative to conventional autologous rib cartilage graft for ear reconstruction for the first time by Reinisch (6). This technique was faced by many arguments like implant fracture, necrosis and failure of healing of the overlying soft tissue due to foreign body reactions to the Medpor implant (5). Many studies were conducted to compare those various techniques specially the Medpor implant and rib cartilage graft but, the superiority of neither of them proved clearly (7).

Aim of the Research :

Evaluation of the outcome of auricular reconstruction in microtia by Medpor implant following tissue expansion.

Research Methods and techniques:

Type of the study:

Prospective randomized controlled clinical trial study.

Study Setting:

The study will be held in the otorhinolaryngology department of Assiut university hospital within duration of three years.

Study subjects: The study will include ten patients

Study tools:

All patients will undergo auricular reconstruction by using a prolonged tissue expansion technique and a Medpor framework at the otorhinolaryngology department of Assiut university hospital following preoperative evaluation which includes:-

* General examination to detect any other medical conditions.
* Complete ENT examination with special emphasis on describing the deformity.
* Audiological and radiological evaluation.
* Full face right and left profile photograph will be taken to be used in the postoperative comparison between the operated auricle and the normal one.

The procedure will be performed in steps:-

* Implantation of the suitable tissue expander in the area of the deformed auricle then after wound healing it will be inflated for three months following removal of postauricular sutures and wound healing during weekly based visits to the department out-patient clinic till it will reach full capacity or even beyond to provide adequate skin for draping the implant.
* The tissue expander will be removed and the Medpor implant "single or double piece" will be applied and covered by the expanded skin flap. All the ten patients will be followed postoperatively for at least six months following the final surgical intervention of the last patient.

Data management and analysis:

Data collection Data will be collected from hospital records about every patient, preoperative, operative and postoperative notes and reports of the physicians.

Computer software Qualitative data will be presented as percentages. Chi-square test (or Fisher's Exact test when applicable) will be used for comparisons between the normal and operated ears regarding qualitative data.

Statistical tests Statistical analysis will be performed with IBM SPSS Statistics Version 20 for Windows.

Ethical Considerations Risk - benefit assessment. Risks and benefits to the participants will be assessed throughout the research in each step. In case of complications as severe infection , tissue necrosis and implant extrusion, the research will be terminated, the case will be considered as failed one and the traditional rib cartilage multistage technique of microtia reconstruction will be performed instead.

Confidentiality (dealing with data and data dissemination should be confidential).

The participants will be reassured before their participation in the research about the confidentiality of their personal and medical data as only research team members will deal with these data. The participants will be reassured that their data will be published in medical journals only after their permission.

Statement describing the research procedure to be given to the participants. Each participant will receive a statement describing the research procedure that will be explained and signed by one of research team members.

Informed consent. Patients or their guardians will be counseled about their participation in the research and the steps of the surgery including application of the tissue expander, the weekly visits for inflation of the expander till it will reach the suitable size permitting enough skin to cover the future device, the possibility of tissue expansion and necrosis and what will be done in such situations. Also they will be counseled about possible complications may occur after each step of the surgery and their important role in assessment of the outcome of the surgery. All the above mentioned points will be written in an informed consent that will be signed by the patient or his guardian.

Other ethical concerns:

- The research should be conducted only by scientifically qualified and trained personnel.

The research will be conducted only by physicians in charge. - The research should be based on relevant pre-clinical investigations in animals.

The research is based on previous similar researches performed on patients published in international medical journals mentioned in the proposal form.

- The consent form must be provided with the proposal Consent of research participation and surgical procedure

I, the undersigned ................, the child's guardian.............. I agree to participate in a research which includes a surgical procedure to repair "microtia" a congenital defect in the ear pinna in two steps. Firstly, tissue expansion by using silicone bag that are placed under the skin behind the ear for a period of about three months, then the second stage is to rebuild the deformed ear pinna by using the Medpor stent. The two stages will be done through a wound behind the deformed ear with knowledge of all the complications received such as failure to reach the optimal shape. Hematoma under the skin or severe infections during any stage of the process, damage or refusal of the stent, severe infections and suppuration of the ear cartilage, which may result in the operation being completely canceled and another surgical intervention will be performed.

References :

1. Tanzer RC. Total reconstruction of the external ear. Plast ReconstrSurg Transplant Bull 1959.
2. Ali K, Trost JG, Truong TA, Harshbarger RJ 3rd. Total Ear Reconstruction Using Porous Polyethylene. Semin Plast Surg.2017.
3. Tjellström A. Osseointegrated implants for replacement of absent or defective ears. Clin Plast Surg 1990.
4. Korus LJ, Wong JN, Wilkes GH. Long-term follow-up of osseointegrated auricular reconstruction. Plast Reconstr Surg2011.
5. Baluch, N., Nagata, S., Park, C., Wilkes, G. H., Reinisch, J., Kasrai, L., & Fisher, D. Auricular reconstruction for microtia: A review of available methods. Plastic surgery (Oakville, Ont.). 2014.
6. Reinisch JF, Lewin S. Ear reconstruction using a porous polyethylene framework and temporoparietal fascia flap. Facial Plast Surg 2009.
7. Constantine KK, Gilmore J, Lee K, Leach J Jr. Comparison of microtia reconstruction outcomes using rib cartilage vs porous polyethylene implant. JAMA Facial Plast Surg. 2014.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral microtia

  * Age not less than six years
  * Non-syndromatic microtia

Exclusion Criteria:

* • Bilateral microtia

  * Age less than six years
  * Syndromatic microtia
  * Previous ear surgery through postauricular incision

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Medpor implant after tissue expansion in treatment of Microtia through comparison with the normal ear regarding skin color, shape, size and patient or relatives satisfaction which will be assessed by likert scale | Three years
  • The research will describe and assess the new technique for reconstruction of microtia by Medpor implant which is a new service not performed in Assiut university that skips the complications of the traditional rib cartilage multistage technique , Also it will assess the degree of patient and family satisfaction. Research on this new service has not been performed in Assiut university.

CONTACTS AND LOCATIONS:
Locations (1):
- AssiutU, Asyut, Egypt